CLINICAL TRIAL: NCT02624882
Title: Impact of Antibiotic Treatment of Group A Streptococcal Blistering Distal Dactylitis in Children
Acronym: TAPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camille JUNG (Other)
Responsible Party: Sponsor-Investigator, Camille JUNG, MD PhD, Centre Hospitalier Intercommunal Creteil
Organization: Centre Hospitalier Intercommunal Creteil (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: TAPPS
Record Dates: First submitted 2015-11-25; First posted 2015-12-09 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Blistering Distal Dactylitis
Keywords: blistering distal dactylitis; Streptococcus pyogenes; antibiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive rapid Group A Streptococcus (GAS) test (Experimental): In case of positive rapid GAS test, patients will be treated by antibiotics: amoxicillin 50mg/kg/d during 10 days or cefpodoxime 8mg/kg/d during 10 days in case of betalactamine allergy
  Interventions: Procedure: Positive rapid GAS test
- Negative rapid GAS test (Active Comparator): If case of negative rapid GAS test, usual care: local antiseptic or surgical intervention
  Interventions: Procedure: Negative rapid GAS test

INTERVENTIONS:
Procedure: Positive rapid GAS test — If TDR positive, the child will be treated with antibiotics alone:
  * Amoxicillin 50mg / kg / day in 2 divided doses for 10 days (maximum dose 3 g / day in 2 divided doses) Or if allergic to penicillins and in the absence of cross-known allergy to cephalosporins
  * Cefpodoxime 8mg / kg / day in 2 divided doses for 10 days (maximum dose 400mg / day in 2 divided doses) J10 A control visit will review all the children included in the study. If the surgeon deems it necessary, the patient will be reviewed in consultation up to three months.
  Arms: Positive rapid Group A Streptococcus (GAS) test
Procedure: Negative rapid GAS test — Usual care
  Arms: Negative rapid GAS test

SUMMARY:
Single-center prospective study to assess the clinical course of group A streptococcal blistering distal dactylitis in children after antibiotic treatment.

DETAILED DESCRIPTION:
Blistering distal dactylitis are very common in children. About 60% are caused by Staphylococcus aureus and some are caused by Group A Streptococcus (GAS) or Streptococcus pyogenes. While these forms have been known for fifty years, few publications are interested in it. Some studies have confirmed that a single antibiotic treatment against the SGA allows the healing of these dactylitis but few surgical teams have adopted this strategy. As all streptococcal infections, they face the risk of acute complications (septicemia, streptococcal toxic shock, etc.) or late (post-streptococcal glomerulonephritis, acute rheumatic fever, etc.). The involvement of the SGA in these dactylitis is easy to demonstrate through the use of rapid GAS test already widely used in other GAS infections (tonsillitis, scarlet fever, streptococcal perianal infections).

This study aims to assess the clinical course of positive GAS test blistering distal dactylitis in children after antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-18 years
* Distal blistering dactylitis collected or not collected
* Positive rapid Group A Streptococcus test
* Informed consent signed by the parents

Exclusion Criteria:

* Subungual or pulp Whitlow
* Children not affiliated to the social security scheme
* Refusal by the parents to participate in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Rate healed blistering distal dactylitis with positive GAS test after 10 days of antibiotherapy directed against streptococcus pyogenes | 10 days
  The main objective of this study is to evaluate the effectiveness of antibiotic treatment only if paronychia subungual child collected or not collected with a in distal blistering dactylitis with positive GAS test

SECONDARY OUTCOMES:
Frequency of distal blistering dactylitis with positive GAS test in children | 18 months
Frequency of collected distal blistering dactylitis with positive GAS test in children | 18 months
Frequency of germs involved in distal blistering dactylitis after pus culture in children | 18 months
Sensitivity of GAS test compared to pus culture | 18 months
  Describe the sensitivity of GAS test in distal blistering dactylitis according to different age groups.
Specificity of GAS test compared to pus culture | 18 months
  Describe the specificity of GAS test in distal blistering dactylitis according to different age groups.
Correlation between GAS test and pus culture in different age groups | 18 months
Number of General anesthesia avoided by use of antibiotics treatment instead of surgical procedure in case of collected distal blistering dactylitis | 18 months
Number of surgical procedures avoided by use of antibiotics treatment instead of surgical procedure in case of collected distal blistering dactylitis | 18 months
Comparison between the cost of antibiotics versus surgical or local treatments of positive GAS test distal blistering dactylitis in children | 18 months
  Evaluate the medical and economic impact of the single antibiotic treatment of distal blistering dactylitis with positive GAS test
Rate of healed collected distal blistering dactylitis with positive GAS test after antibiotic treatment | 18 months
Number of Nail dystrophy at 3 months of follow-up | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Camille Jung, MD, PhD, Principal Investigator — CHIC Créteil
Locations (1):
- CHI Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No